CLINICAL TRIAL: NCT07331077
Title: Movement and Memory After Breast Cancer: The MAMA Trial
Brief Title: A Physical Activity Program Compared to Health Education for Improving Memory and Attention in Hispanic Women With Newly-Diagnosed Stage I-IIIa Breast Cancer, MAMA Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-007121; NCI-2025-08551 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 25-007121 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2025-12-09; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Cancer-related Cognitive Dysfunction
MeSH Terms: interventions — Accelerometry; Exercise; Interviews as Topic; Mental Status and Dementia Tests; Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (walking program) (Experimental): Patients participate in walking sessions over 60-75 minutes per week in weeks 1-2, 70-90 minutes per week in weeks 3-4, 90-120 minutes per week in weeks 5-8, 120-135 minutes per week in weeks 9-12, 135-150 minutes per week in weeks 13-16, and 150+ minutes per week in weeks 17-24. Patients also undergo fMRI throughout the trial.
  Interventions: Procedure: Accelerometry; Other: Aerobic Exercise; Other: Electronic Health Record Review; Procedure: Functional Magnetic Resonance Imaging; Other: Gait Assessment Test; Other: Interview; Other: Neurocognitive Assessment; Other: Physical Performance Testing; Other: Questionnaire Administration
- Arm B (health education) (Active Comparator): Patients receive health education including monthly classes/webinars for up to 9 sessions and informational materials (PDFs, videos, podcasts, and/or subscription to Mayo Clinic Health Letter). Patients also undergo fMRI throughout the trial.
  Interventions: Procedure: Accelerometry; Other: Electronic Health Record Review; Procedure: Functional Magnetic Resonance Imaging; Other: Gait Assessment Test; Behavioral: Health Education; Other: Neurocognitive Assessment; Other: Physical Performance Testing; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Accelerometry — Ancillary studies
Other: Aerobic Exercise — Participate in walking program
  Other Names: Aerobic Activity
  Arms: Arm A (walking program)
Other: Electronic Health Record Review — Ancillary studies
Procedure: Functional Magnetic Resonance Imaging — Undergo fMRI
  Other Names: fMRI; Functional MRI
Other: Gait Assessment Test — Ancillary studies
Behavioral: Health Education — Receive health education
  Arms: Arm B (health education)
Other: Interview — Ancillary studies
  Arms: Arm A (walking program)
Other: Neurocognitive Assessment — Ancillary studies
Other: Physical Performance Testing — Ancillary studies
  Other Names: Physical Fitness Testing; Physical Function Testing
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial compares a physical activity program to a health education program for improving memory and attention in Hispanic women who are 50 years of age or older and are newly-diagnosed with stage I-IIIa breast cancer. Compared to non-Hispanic White breast cancer survivors (BCS), Hispanic BCS report greater depressive symptoms, emotional distress, anxiety, fear of recurrence, pain, fatigue, and financial toxicity, in addition to more cancer-related psychosocial needs and lower quality of life and social well-being. Cancer-associated cognitive decline (CACD) is a related symptom that has gained increasing attention in clinical research. Based on disparities in other outcomes, it is likely that Hispanic BCS also experience greater CACD than non-Hispanic White BCS, but interventions targeting CACD in Hispanic BCS are non-existent and critically needed. The benefits of aerobic exercise among BCS are well documented and include improvement in health outcomes that are associated with cognitive function including fatigue, anxiety, depression, and sleep. A physical activity program that includes aerobic exercise may be more effective than simple health education for improving cognitive functions like memory and attention in Hispanic women who are 50 years of age or older and are newly-diagnosed with stage I-IIIa breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION: Age >= 50 years at time of pre-registration visit according to participant report and/or clinical determination
* PRE-REGISTRATION: Self-identifies as Hispanic (any race)
* PRE-REGISTRATION: First time, primary diagnosis of Stage I-IIIa breast cancer according to participant report and/or clinical determination
* PRE-REGISTRATION: Post-surgery and completed primary adjuvant treatment (i.e., surgery, chemotherapy, and/or radiation therapy) 3-36 months prior to preregistration according to participant report and/or clinical determination
* PRE-REGISTRATION: Sedentary except for casual lifestyle recreation, self-reporting no more than 90 minutes per week of moderate-intensity aerobic exercise within the last 6 months
* PRE-REGISTRATION: Self-reported ability to complete assessments by themselves or with assistance
* REGISTRATION: Age >= 50 years or older as confirmed via clinical determination
* REGISTRATION: Self-identifies as Hispanic (any race)
* REGISTRATION: Able to provide medical record release to confirm eligibility
* REGISTRATION: First time, primary diagnosis of Stage I-IIIa breast cancer as confirmed via clinical determination
* REGISTRATION: Post-surgery and completed primary treatment (i.e., surgery, chemotherapy, and/or radiation therapy) 3-36 months prior to pre-registration as confirmed via clinical determination
* REGISTRATION: No evidence of possible cognitive impairment as assessed using the Telephone Interview of Cognitive status (13-item modified version) (TICS-M; score >= 21)
* REGISTRATION: Receive physician's clearance to participate in an exercise program

  * NOTE: Individuals with conditions/diagnoses deemed important by the primary investigator will be required to provide clearance for exercise from their cardiologist. Example conditions include:

    * History of major multiple myocardial infarctions (MI)
    * Recent electrocardiogram (ECG) changes or recent MI
    * Resting or unstable angina
    * Significant multivessel coronary occlusion (>= 70%) on angiography
    * Uncontrolled and/or serious arrhythmias
    * 3rd degree heart block
    * Acute congestive heart failure or ejection fraction < 30%
* REGISTRATION: Ability to complete assessments by themselves or with assistance
* REGISTRATION: Agree to be randomized

Exclusion Criteria:

* PRE-REGISTRATION: Stage 0 breast cancer diagnosis OR metastatic disease
* PRE-REGISTRATION: Currently receiving or < 3 months since receiving chemotherapy or radiation therapy for cancer, or greater than 36 months post primary treatment
* PRE-REGISTRATION: Planned surgery during the intervention period
* PRE-REGISTRATION: Secondary cancer diagnosis (excluding non-invasive skin cancers, carcinoma-in-situ for any cancer)
* PRE-REGISTRATION: Unable to regularly attend the study locations for intervention sessions and data collection
* PRE-REGISTRATION: Unwilling to return to enrolling institution for follow-up
* PRE-REGISTRATION: Self-reported inability to walk without assistance or devices
* PRE-REGISTRATION: Self-reported pregnancy
* REGISTRATION: History of stroke, transient ischemic attack, other neurological disorders, or brain surgery involving tissue removal as confirmed via clinical determination
* REGISTRATION: Clinically significant TICS-M score (< 21) during baseline procedures
* REGISTRATION: Not able to provide physician re-clearance for exercise if required based upon clinically significant baseline exercise test (as determined by ECG and blood pressure monitoring)
* REGISTRATION: Contraindications to functional magnetic resonance imaging (fMRI) in accordance with the Mayo Clinic Department of Radiology safety protocols
* REGISTRATION: Clinically significant magnetic resonance imaging (MRI) scan as determined by physician review in which the following is advised via radiologist overread: remarkable/abnormal limited diagnostic brain image with recommended medical follow-up
* REGISTRATION: Enrolled in another physical activity program
* REGISTRATION: Unable to walk without assistance or devices
* REGISTRATION: Unwilling to complete study requirements
* REGISTRATION: Unwilling to be randomized to the exercise group or health education group
* REGISTRATION: Unable to regularly attend study locations for intervention sessions and data collection
* REGISTRATION: Unwilling to return to enrolling institution for follow-up
* REGISTRATION: Unable to complete the study in English or Spanish
* REGISTRATION: Self-reported pregnancy

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in inhibitory control | Baseline to post-intervention (month 6)
  Change in interference score on Stroop task, with positive values indicating greater inhibitory control
Change in cognitive flexibility | Baseline to post-intervention (month 6)
  Change in accuracy on Shifting Attention task, with higher values indicating greater cognitive flexibility
Change in executive function processing | Baseline to post-intervention (month 6)
  Change in reaction time on Shifting Attention task, with lower values indicating greater cognitive flexibility
Change in short-term memory | Baseline to post-intervention (month 6)
  Change in accuracy on Visual Memory task, with higher accuracy indicating greater short-term memory
Change in verbal memory | Baseline to post-intervention (month 6)
  Change in number recalled on Hopkins Verbal Learning task, with higher values indicating greater verbal memory
Change in working memory | Baseline to post-intervention (month 6)
  Change in reaction time the 4-part Continuous Performance task, with lower values indicating greater working memory
Change in processing speed | Baseline to post-intervention (month 6)
  Change in reaction time on Symbol Digit Coding task, with lower values indicating greater processing speed
Change in attention | Baseline to post-intervention (month 6)
  Change in choice reaction time on Continuous Performance task, with lower values indicating greater sustained attention
Change in brain volume | Baseline to post-intervention (month 6)
  Change in mean cortical thickness of brain regions of interest as measured by an anatomic MRI brain scan
Change in white matter integrity | Baseline to post-intervention (month 6)
  Change in fractional anisotropy as measured by diffusion MRI.
Change in resting state functional connectivity | Baseline to post-intervention (month 6)
  Change in within-network pairwise correlation estimates as measured using a multiband echo planar imaging (mb-EPI) functional MRI sequence
Change in self-reported cognitive function - FACT-Cog | Baseline to post-intervention (month 6)
  The perceived cognitive impairments subscale of the Functional Assessment in Cancer Therapy - Cognition (FACT-Cog) will be used to measure self-reported cognition. Scores range from 0-72, with higher scores indicating better cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Diane K. Ehlers, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials